CLINICAL TRIAL: NCT02311088
Title: Trial of Caffeine to Alleviate Dyspnea Related to Ticagrelor - A Double-blinded, Placebo-controlled, Randomized, Multicenter, Development Phase II Study
Brief Title: Trial of Caffeine to Alleviate Dyspnea Related to Ticagrelor
Acronym: TROCADERO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Too low enrolment rate
Sponsor: Uppsala University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U-2013-007; 2013-004412-22 (EudraCT Number)
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Caffeine (Experimental): Caffeine capsules. 200 mg twice daily orally for 7-10 days.
  Interventions: Drug: Caffeine
- Placebo (Placebo Comparator): Matching placebo capsules twice daily orally for 7-10 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Caffeine
  Arms: Caffeine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Ticagrelor treatment is associated with increased rates of dyspnea, where previous studies have implied a possible role of adenosine. The purpose of this study is to determine if the caffeine-antagonist is effective in reducing dyspnea related to ticagrelor.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Recent acute coronary syndrome with ongoing ticagrelor treatment
* Stabilized clinical condition with no plans of additional revascularization
* Dyspnea with onset after start of ticagrelor treatment
* Willingness to abstain from caffeine intake (e.g. coffee, tea, cola-type beverages; other foods, nutritional supplements or medications containing caffeine) for the duration of the study
* Provision of signed informed consent form

Exclusion Criteria:

* Chronic obstructive pulmonary disease, asthma or other known pulmonary disease requiring daily medical therapy
* Obstructive sleep apnea syndrome requiring therapy
* Ongoing signs and symptoms of heart failure*, or evidence of moderately to severely reduced left ventricular (LV) function
* Renal failure, glomerular filtration rate (GFR) <30 or on dialysis
* Pregnancy or lactation
* Known allergy to ticagrelor, or caffeine, or known intolerance of caffeine
* Ongoing treatment with any of the following: quinolone antibiotics, fluvoxamine, phenylpropanolamine, carbamazepine, clozapine, lithium, non-steroidal anti-inflammatory drugs (NSAIDs); or any drug containing theophylline or caffeine.
* Any condition that seriously increases the risk of non-compliance or loss of follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Visual analog scale area under the curve (VAS-AUC) for dyspnea | 7-10 days

SECONDARY OUTCOMES:
High on-treatment platelet reactivity by VerifyNow | 7-10 days
Change in dyspnea by 7-point Likert scale | 7-10 days

CONTACTS AND LOCATIONS:
Overall Officials: Stefan K James, MD, PhD, Principal Investigator — Uppsala University
Locations (9):
- Sweden (9):
  - Dept of Cardiology, Mälarsjukhuset hospital, Eskilstuna
  - Dept. of Cardiology, Falu hospital, Falun
  - Dept of Cardiology, Gävle Hospital, Gävle
  - Dept of Cardiology, Östra hospital, Gothenburg
  - Dept. of Cardiology, Linköping University Hospital, Linköping
  - Dept of Cardiology, Skåne University Hospital, Lund
  - Dept. of Cardiology, Danderyd hospital, Stockholm
  - Dept of Cardiology, Umeå University Hospital, Umeå
  - Dept of Cardiology, Uppsala University Hospital, Uppsala

REFERENCES:
- [Derived] Lindholm D, James S, Andersson J, Braun OO, Heller S, Henriksson P, Lauermann J, Ohagen P, Varenhorst C. Caffeine and incidence of dyspnea in patients treated with ticagrelor. Am Heart J. 2018 Jun;200:141-143. doi: 10.1016/j.ahj.2018.02.011. Epub 2018 Feb 16. No abstract available. PMID 29898843